CLINICAL TRIAL: NCT00089037
Title: A Phase I/II Study of Sirolimus in Addition to Tacrolimus and Methotrexate for the Prevention of Acute-Graft-Versus-Host Disease in Patients Undergoing Hematopoietic Stem Cell Transplantation From Unrelated Donors
Brief Title: Sirolimus, Tacrolimus, and Methotrexate in Preventing Acute Graft-Versus-Host Disease in Patients With Hematologic Cancer Who Are Undergoing Donor Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Kiem, Hans-Peter, Fred Hutchinson Cancer Research Center
Masking: None | Purpose: Supportive Care
Other Study IDs: 1811.00; FHCRC-1811.00; CDR0000378004 (Registry Identifier: PDQ)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; accelerated phase chronic myelogenous leukemia; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; de novo myelodysplastic syndromes; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; noncontiguous stage II adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; childhood chronic myelogenous leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; recurrent/refractory childhood Hodgkin lymphoma; juvenile myelomonocytic leukemia; splenic marginal zone lymphoma; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory cytopenia with multilineage dysplasia; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Dendritic Cell Sarcoma, Interdigitating; Recurrence; Leukemia, Myelomonocytic, Juvenile; Lymphoma, T-Cell, Cutaneous | interventions — Methotrexate; Sirolimus; Tacrolimus

INTERVENTIONS:
Drug: methotrexate
Drug: sirolimus
Drug: tacrolimus

SUMMARY:
RATIONALE: Sirolimus, tacrolimus, and methotrexate may be effective in preventing acute graft-versus-host disease in patients who are undergoing donor stem cell transplantation.

PURPOSE: This phase I/II trial is studying the side effects of sirolimus when given together with tacrolimus and methotrexate and to see how well they work in preventing acute graft-versus-host disease in patients who are undergoing donor stem cell transplantation for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and efficacy of sirolimus when administered with tacrolimus and methotrexate for the prevention of acute graft-versus-host disease (GVHD) in patients with hematological malignancies undergoing hematopoietic stem cell transplantation from unrelated donors.

Secondary

* Determine the absorption and pharmacokinetics of sirolimus in patients treated with this regimen.
* Correlate sirolimus blood concentration with prevention of GVHD or toxicity in patients treated with this regimen.
* Determine the severity of post-transplantation mucositis in patients treated with this regimen.

OUTLINE: This is a nonrandomized, open-label, pilot study.

Patients receive oral sirolimus once daily on days -3 to 175 and tacrolimus IV continuously beginning on day -3 and continuing until the patient is able to tolerate food and then orally twice daily until day 175. Patients also receive methotrexate IV on days 1, 3, 6, and 11. Treatment continues in the absence of acute graft-vs-host disease or unacceptable toxicity.

Patients are followed for 5 years.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hematological malignancy

  * No chronic phase chronic myelogenous leukemia, de novo acute leukemia in first remission, or myelodysplastic syndromes with refractory anemia
* Scheduled for hematopoietic stem cell transplantation from unrelated donors
* Currently receiving conditioning regimen comprising cyclosporine and total body radiotherapy (1,200 to 1,350 cGy) or busulfan and cyclosporine
* Donor must be typed to the highest level of resolution

  * One single non-serologic disparity for A, B, or C alleles allowed provided the disparity is within the third or fourth digit of the allele
  * No mismatch at DRB1 or DQB1

PATIENT CHARACTERISTICS:

Age

* Per primary treatment protocol

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* SGOT and SGPT ≤ 2.0 times upper limit of normal
* Bilirubin normal
* Hepatitis B and C virus negative

Renal

* Creatinine clearance ≥ 70 mL/min

Cardiovascular

* No cardiac insufficiency requiring treatment
* No coronary artery disease

Pulmonary

* No acute pulmonary infection by chest x-ray
* No severe hypoxemia with pO_2 < 70 mm Hg AND DLCO < 70% of predicted
* No mild hypoxemia with pO_2 < 80 mm Hg AND DLCO < 60% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* HIV negative
* No active systemic infection
* No known hypersensitivity to macrolide antibiotics (e.g., erythromycin, azithromycin, or clarithromycin)
* No prior intolerance or unresponsiveness to sirolimus

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No concurrent T-cell depleted transplantations

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* No concurrent grapefruit juice
* No concurrent voriconazole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Kiem, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States